CLINICAL TRIAL: NCT04461964
Title: Single Center, Prospective Study of the MvIGS Spine Navigation System in Posterior Fusion Utilizing Pedicle Screw Fixation
Brief Title: Effects of a Spine Navigation System on Op-time and Radiation Exposure
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: funding for the study has stopped
Sponsor: NYU Langone Health (Other)
Collaborators: 7D Surgical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-01201
Record Dates: First submitted 2020-06-30; First posted 2020-07-08 (Actual); Last update posted 2022-06-13 (Actual); Status verified 2022-06

CONDITIONS: Spinal Stenosis; Scoliosis; Spondylolisthesis
MeSH Terms: conditions — Spinal Stenosis; Scoliosis; Spondylolisthesis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment group (Experimental): Eligible participants will be identified by their treating physician and referred to the study research coordinator for enrollment. NYU standard practice in relation to pre-operative and intra-operative imaging studies will be explained. The role of the MvIGS system in this study will then also be explained. In each subject, they will perform posterior instrumentation utilizing the MvIGS spine navigation system for pedicle screw guidance and record data for intraoperative study endpoints
  Interventions: Device: Machine-vision Image Guided Surgery (MvIGS) spine navigation system.

INTERVENTIONS:
Device: Machine-vision Image Guided Surgery (MvIGS) spine navigation system. — The intended use of the MvIGS navigation system is to provide high quality intraoperative imaging with no radiation exposure. Use of the proprietary integrated surgical light with embedded tracking technology and Flash™ registration allows for continuous and direct visualization of the surgical field. The MvIGS system is exempt from IDE regulations as the device cleared Premarket Notification FDA-510(k) (K162375). The device includes:
  * A single mobile cart with a boom arm and an integrated surgical light with embedded tracking technology (P/N 10-0001);
  * Proprietary imaging software (P/N 60-0007); and,
  * Kit of tacked surgical instruments including a spine reference clamp, awl tip, pedicle probe (P/N 11-0006).

SUMMARY:
The goal of this study is to prospectively collect information about the operative time and intraoperative radiation experienced by patients undergoing posterior spinal fusion procedures guided by the MvIGS spine navigation system.

DETAILED DESCRIPTION:
This is a single-center, prospective case series to assess the use of the Machine-vision Image Guided Surgery (MvIGS) spine navigation system for treatment of spinal stenosis, scoliosis, and spondylolisthesis that requires fusion. This is a single-arm, open-label study. All participants will undergo their single and multi-level posterior spine fusion surgery using bilateral pedicle screw instrumentation under MvIGS intraoperative navigation guidance.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of spinal stenosis of the lumbar spine with degenerative spondylolisthesis, all grades, and planning to undergo surgical fusion;
* Skeletally mature adults between the ages of 18-85 years at the time of surgery;
* Has completed at least 6 months of conservative therapy for degenerative diagnosis, if appropriate; and,
* Personally signed and dated an informed consent document prior to any study-related procedures, indicating that the patient has been informed of all pertinent aspects of the study.

Exclusion Criteria:

* History of malignancy, craniocervical junction pathology, cervical and thoracic locations, and/or previous lumbar operation;
* Significant peripheral neuropathy or acute denervation secondary to radiculopathy, caused by conditions other than spinal stenosis;
* Significant peripheral vascular disease (defined as diminished dorsalis pedis or tibial pulses);
* Morbid obesity, defined as BMI > 40 kg/m2;
* Active systemic or local infection;
* Active hepatitis (defined as receiving medical treatment within two years);
* Immunocompromised, such as but not limited to being diagnosed with Acquired Immunodeficiency Syndrome (AIDS), HIV infection, Severe Combined Immunodeficiency Syndrome, or Thymic Hypoplasia;
* Insulin-dependent diabetes mellitus or any other medical condition(s) that would represent a significant increase in surgical risk or interfere with normal healing;
* Immunologically suppressed, or has received systemic steroids, excluding nasal steroids, at any dose daily for > 1 month within last 12 months;
* History of Paget's disease, osteomalacia, or any other metabolic bone disease;
* Involved in study of another investigational product that may affect outcome;
* Women who are pregnant, lactating or anticipate becoming pregnant within 24 months post-surgery;
* Non-English speaking;
* Patients who are incarcerated;
* Worker's compensation cases; or,
* Patients involved in active litigation relating to his/her spinal condition.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-07 (Estimated); Primary Completion 2023-02 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Total length of operative time | Visit 1 Day 1
  The aim is to reduce operative time. Operative time will be determined by the official recorded operative notes.

SECONDARY OUTCOMES:
Length of time to register images | Visit 1 Day 1
  Aim: To reduce time for registration of reference images Measured: Seconds
Length of time to place all screws | Visit 1 Day 1
  Aim: To reduce the time for screw placement Measured: Minutes
Estimated blood loss (EBL) | Visit 1 Day 1
  Aim: To reduce the EBL of each case Measured: Millilitres (mL)
Dose of intraoperative ionizing radiation | Visit 1 Day 1
  Aim: To reduce intraoperative ionizing radiation Measured: Total amount of the radiation dose in millisievert (mSv)
Screw placement accuracy | Visit 1 Day 1
  Aim: To improve screw placement accuracy Measured: Graded using radiographic classification and clinical revision rate
incidence of intraoperative complications | Visit 1 Day 1
  Aim: To decrease the incidence of intraoperative complications Measured: Number of reported complications
Time to ambulation | Post operative hospital visit (Day 1-10)
  Aim: To reduce time to ambulation Measured: Days
Time to hospital discharge after surgery | Post operative hospital visit (Day 1-10)
  Aim: To reduce hospital length of stay Measured: Days

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey A Goldstein, MD, Principal Investigator — NYU Langone Health

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data. Upon reasonable request. Requests should be directed to Jeffrey.goldstein@nyulangone.org . To gain access, data requestors will need to sign a data access agreement.